CLINICAL TRIAL: NCT01666028
Title: An Open-label, Three-centre, Randomised, Two-period Crossover Study to Assess the Safety, Efficacy and Utility of Automated Closed-loop Glucose Control in Comparison With Continuous Subcutaneous Insulin Infusion Combined With Continuous Glucose Monitoring in Adults With Type 1 Diabetes - A Combined Clinical Research Facility and Home Study
Brief Title: Short Term Closed-loop Glucose Control in Adults With Type 1 Diabetes
Acronym: AP@home02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Profil Institut für Stoffwechselforschung GmbH (Industry); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Principal Research Associate, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AP@home02
Record Dates: First submitted 2012-08-09; First posted 2012-08-16 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Closed Loop glucose control; Artificial Pancreas; CSII; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed Loop Glucose control (Experimental): Subject's glucose level is controlled by the automated closed loop glucose control system
  Interventions: Device: FlorenceD or similar closed loop glucose control system
- CSII with real-time CGM (Active Comparator): Subject glucose level controlled by usual insulin pump therapy in conjunction with real time continuous glucose monitoring (CGM)
  Interventions: Device: CSII with real-time CGM

INTERVENTIONS:
Device: FlorenceD or similar closed loop glucose control system — Subject's glucose level will be controlled by the FlorenceD or similar automated closed loop glucose control system. The system comprises of FreeStyle Navigator® Continuous Glucose Monitoring (CGM) System (Abbott Diabetes Care, Alameda, CA, USA), Dana R Diabecare subcutaneous insulin infusion pump (Sooil Corp. Seoul, South Korea)or similar insulin pump, and MPC-based glucose control algorithm running on a portable computer.
  Arms: Closed Loop Glucose control
Device: CSII with real-time CGM — Subject glucose level controlled by usual insulin pump therapy in conjunction with real time continuous glucose monitoring (CGM)
  Arms: CSII with real-time CGM

SUMMARY:
The main objective of this study is to determine the feasibility, efficacy and safety of automated closed-loop glucose control in the home setting over a short term period. The data and experienced gained from this study will be utilised in planning future home studies.

This is an open-label, three centre, randomised, crossover design, involving two, 8 day (first day in the clinical research facility and seven days at home) study periods during which glucose levels will be controlled either by an automated closed-loop system or by subjects usual insulin pump therapy in random order. A total of up to 24 adults (aiming for 18 completed subjects) aged 18 years and older with T1D on insulin pump therapy will be recruited through diabetes clinics and other established methods in participating centres.

Subjects will receive appropriate training in the safe use of closed-loop insulin delivery system. During the 24 hour in-patient stay subjects will be encouraged to mimic their usual day and will be allowed to walk inside hospital premises. Subjects will be advised to discontinue automated closed-loop insulin delivery and follow their usual insulin pump therapy for periods of strenuous exercise during the 7 day home study phase.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM (adjusted for potential over-estimation) during home stay. Secondary outcomes are the time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics, and for the stay at the clinical research facility, time spent in the target range, above and below the target range as measured by plasma glucose.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has type 1 diabetes as defined by WHO
2. The subject is 18 years of age or older
3. The subject will have been on an insulin pump for at least 3 months currently using insulin Aspart, with good knowledge of insulin self-adjustment including carbohydrate counting
4. HbA1c ≤ 10 % based on analysis from local laboratory
5. The subject is willing to perform regular finger-prick blood glucose monitoring, with at least 6 measurements per day during the 7 day home phase of the study
6. The subject is willing to wear closed-loop system at home and at work place
7. The subject is willing to follow study specific instructions
8. The subject is literate in English
9. Female subjects of child bearing age should be on effective contraception and must have a negative urine-HCG pregnancy test at screening. In addition in Germany, women of childbearing potential must use a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e. less than 1% per year) and must use two independent methods of contraception, e.g. diaphragm and spermicide-coated condom.

Exclusion Criteria:

1. Non-type 1 diabetes mellitus
2. Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
3. Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
4. Known or suspected allergy against insulin
5. Subjects with clinically significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
6. Significantly reduced hypoglycaemia awareness as judged by the investigator
7. Total daily insulin dose more than 2 IU/kg/day
8. Subject is pregnant or breast feeding or planning pregnancy in near future (within next 3 months)
9. Severe visual impairment
10. Severe hearing impairment
11. Subjects using implanted internal pacemaker
12. Lack of reliable telephone facility for contact

Additional exclusion criteria specific for Austria and Germany

1. Positive results on urine drug screen (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
2. Positive alcohol breath test.

Additional exclusion criteria specific for Germany only

Positive reaction to any of the following tests: hepatitis B surface (HBs) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus (HIV) 1 antibodies, anti-HIV2 antibodies

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring (CGM) adjusted for sensor error. | 7 day home study period

SECONDARY OUTCOMES:
Time spent above and below the target glucose (3.9 to 10.0 mmol/l) based on continuous subcutaneous glucose monitoring (CGM) | 7 day home study period
Average and standard deviation glucose levels based on continuous subcutaneous glucose monitoring | 7 day home study period
The time with glucose levels < 3.5 mmol/l and <2.8 mmol/l based on continuous subcutaneous glucose monitoring | 7 Day home study period
The time with glucose levels in the significant hyperglycaemia, as based on continuous subcutaneous glucose monitoring (glucose levels > 16.7 mmol/l) | 7 day home study period
Low Blood Glucose Index (LBGI) based on continuous subcutaneous glucose monitoring | 7 day Home study period
During 24 hour in-patient stay - Same glucose metrics as during 7 day home stay but calculated based on continuous subcutaneous glucose monitoring (CGM) and plasma glucose measurements. | 24 hours
Number of episodes of hypoglycaemia, severe hypoglycaemia as well as nature and severity of any other adverse events. | 8 days

OTHER OUTCOMES:
Duration of use of the closed-loop system at home. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Evans, FRCP (UK) MD, Principal Investigator — University of Cambridge; Sabine Arnolds, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH; Thomas Pieber, MD, Principal Investigator — Medical University of Graz; Roman Hovorka, PhD, Study Director — University of Cambridge
Locations (3):
- Medical University of Graz, Graz, Austria
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357
- [Background] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665
- [Derived] Thabit H, Leelarathna L, Wilinska ME, Elleri D, Allen JM, Lubina-Solomon A, Walkinshaw E, Stadler M, Choudhary P, Mader JK, Dellweg S, Benesch C, Pieber TR, Arnolds S, Heller SR, Amiel SA, Dunger D, Evans ML, Hovorka R. Accuracy of Continuous Glucose Monitoring During Three Closed-Loop Home Studies Under Free-Living Conditions. Diabetes Technol Ther. 2015 Nov;17(11):801-7. doi: 10.1089/dia.2015.0062. Epub 2015 Aug 4. PMID 26241693
- [Derived] Leelarathna L, Dellweg S, Mader JK, Allen JM, Benesch C, Doll W, Ellmerer M, Hartnell S, Heinemann L, Kojzar H, Michalewski L, Nodale M, Thabit H, Wilinska ME, Pieber TR, Arnolds S, Evans ML, Hovorka R; AP@home Consortium. Day and night home closed-loop insulin delivery in adults with type 1 diabetes: three-center randomized crossover study. Diabetes Care. 2014 Jul;37(7):1931-7. doi: 10.2337/dc13-2911. PMID 24963110